CLINICAL TRIAL: NCT01228279
Title: Effects of Non-Glucose-Based Peritoneal Dialysis Solution "EXTRANEAL" on Changes in Leptin Levels and Sympathetic Activity Induced by Conventional Glucose-Based Dialysate "DIANEAL" in Patients on Peritoneal Dialysis
Brief Title: Sympathetic Activity in Patients With End-stage Renal Disease on Peritoneal Dialysis
Acronym: SAPD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Heart and Stroke Foundation of Ontario (Other)
Responsible Party: Principal Investigator, Dr. Marcel Ruzicka, Dr. Marcel Ruzicka, Ottawa Hospital Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NA6951
Record Dates: First submitted 2010-10-13; First posted 2010-10-26 (Estimated); Last update posted 2021-03-15 (Actual); Status verified 2021-03

CONDITIONS: End-stage Renal Disease (ESRD); Kidney Disease
Keywords: Peritoneal Dialysis; Dialysis Solutions; Artificial Kidney; Renal Replacement Therapy; Renal Dialysis; Sympathetic Nervous System; Leptin; Icodextrin
MeSH Terms: conditions — Kidney Failure, Chronic; Kidney Diseases | interventions — Icodextrin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DIANEAL (Active Comparator): One group of patients will start peritoneal dialysis with the glucose-based solution (DIANEAL) for 6 weeks, then will continue with the same type of solution for another 12 weeks.
  Interventions: Other: DIANEAL
- EXTRANEAL (Active Comparator): The other group of patients will start peritoneal dialysis with the glucose-based solution (DIANEAL) for 6 weeks, then will continue with DIANEAL solution during the day and the non-glucose-based solution, EXTRANEAL, during the night
  Interventions: Other: EXTRANEAL

INTERVENTIONS:
Other: DIANEAL — Weeks 1 to 6 (6 weeks):
  * CAPD (Continuous Ambulatory Peritoneal Dialysis)patients will receive three 4-6 hour dwells of DIANEAL during the day and one 8-10-hour dwell of DIANEAL during the night
  * CCPD (Continuous Cycler Peritoneal Dialysis)patients will receive one-two 4-6 hour dwells of DIANEAL during the day and three to seven 2-4-hour dwells of DIANEAL during the night
  Weeks 7 to 18 (12 weeks):
  *same regimen as weeks 1 to 6, for both CAPD and CCPD patients
  Other Names: Dextrose-based PD solution
  Arms: DIANEAL
Other: EXTRANEAL — Weeks 1 to 6 (6 weeks):
  * CAPD (Continuous Ambulatory Peritoneal Dialysis)patients will receive three 4-6 hour dwells of DIANEAL during the day and one 8-10-hour dwell of DIANEAL during the night
  * CCPD (Continuous Cycler Peritoneal Dialysis)patients will receive one-two 8-12-hour dwells of DIANEAL during the day and three to seven 2-4-hour dwells of DIANEAL during the night
  Weeks 7 to 18 (12 weeks):
  * CAPD (Continuous Ambulatory Peritoneal Dialysis)patients will receive three 4-6 hour dwells of DIANEAL during the day and one 8-10-hour dwell of EXTRANEAL during the night
  * CCPD (Continuous Cycler Peritoneal Dialysis)patients will receive one-two 8-12-hour dwells of DIANEAL during the day and one 8-12-hour dwell of EXTRANEAL during the night
  Other Names: Icodextrin-based PD solution
  Arms: EXTRANEAL

SUMMARY:
Hypothesis:

Patients starting peritoneal dialysis with a glucose-based regimen have high sympathetic activity in response to an increase in leptin and insulin. Converting patients from a regimen of only glucose containing dialysate to a regimen with non-glucose-based solution, icodextrin, will reduce the insulin and leptin levels and will reverse dialysis-induced increases in sympathetic activity.

DETAILED DESCRIPTION:
Cardiovascular mortality remains higher among patients treated with peritoneal dialysis as compared to patients treated with hemodialysis. Sympathetic hyperactivity is considered a significant emerging risk factor for cardiovascular mortality among patients with ESRD (End-Stage Renal Disease). Sympathetic activity, via its hemodynamic effects and trophic effects, and in interaction with RAAS (Renin Angiotensin Aldosterone System), does play a major role in cardiac and vascular remodelling, development of LVH and vascular hypertrophy, as well as progression to CHF. Glucose-based dialysate induces hyperinsulinemia and hyperleptinemia. We propose that hyperleptinemia induced by glucose-based peritoneal solution is a significant contributing factor to sympathetic hyperactivity in ESRD patients treated with PD, and could be prevented by non-glucose-based PD solution such as icodextrin-based.

Adult patients with ESRD starting PD as their first renal replacement therapy modality will be studied. Patients will be recruited 1-3 weeks prior to starting PD treatment. At baseline, specific studies for microneurography (MSNA), fasting plasma insulin, leptin, catecholamines and brain natriuretic peptide (BNP) will be performed. EKG will be recorded and digitized for further assessment of heart rate variability using power spectral analysis. Extracellular fluid volume status will be assessed by bioelectrical impedance. Central vascular volume will be assessed from inferior vena cava (IVC) by heart ultrasound. Consequently 24-h ambulatory blood pressure monitoring(ABPM)and a 24-h urine collection for urea clearance and creatinine clearance will be done.

All participants into the study will receive a PD treatment for 6 weeks with standard glucose-based PD solution Dianeal. The specific studies are repeated at 6 weeks.Then, patients will be randomized to one of the two groups (arms). One group will continue with Dianeal PD solution for another 12 weeks. The other group will receive Dianeal during the day and Extraneal, icodextrin or non-glucose based solution, during the night only, for the next 12 weeks. The specific studies are repeated at 12 weeks after randomization (18 weeks of PD treatment).

ELIGIBILITY:
Inclusion Criteria:

* Adult (age 18 years and older)
* Patients with end-stage renal disease(ESRD)/chronic kidney disease(CKD)stage 5

Exclusion Criteria:

* Diabetes Mellitus
* Acute coronary syndrome in the past 6 months
* Cardiac arrhythmias (2nd and 3rd degree heart block or premature ventricular complexes in Lown classes 4 or 5)
* Symptoms suggestive of obstructive or central sleep apnea (with a score of > 10 on Epworth sleepiness scale)
* Patients taking Clonidine
* Body mass index (BMI) > 34
* Patients unable to give consent
* Pregnant women
* Patients with leg injury involving nerve damage
* Patients taking anticoagulant medication
* Patients with significant bleeding disorder or liver disorder
* Hemoglobin <1.05 g/dl at the time of initiation of therapy
* patients with unilateral or bilateral nephrectomy
* Planned kidney transplant in the next 4 months
* Life expectancy under 6 months
* Oliguria (urine output less than 400 ml per day)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2007-07 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Changes in muscle sympathetic nerve activity(MSNA) | 6 weeks on PD and 18 weeks on PD
  Muscle sympathetic nerve activity(MSNA) is measured by microneurography at
  * baseline (before starting peritoneal dialysis)
  * 6 weeks of PD
  * 18 weeks of PD(12 weeks after randomization)
  MSNA increases on a glucose-based dialysis regimen and may decrease by adding non-glucose-based solution
Changes in leptin levels | 6 weeks on PD and 18 weeks on PD
  Plasma leptin increases on a glucose-based peritoneal dialysis regimen and may decrease by adding non-glucose-based solution to the dialysis regimen

SECONDARY OUTCOMES:
Changes in blood pressure as assessed from 24-hour ambulatory blood pressure monitor (ABPM) | 6 weeks on PD and 18 weeks on PD
  Blood pressure will be assessed with 24-hour ABPM at baseline, 6 weeks on PD and 18 weeks after starting peritoneal dilaysis. Summary measures of each day and night period include average systolic and diastolic BP as well as % nocturnal dipping. These summary measures can predict cardiovascular events more accurately than casual BP measures
Changes in extracellular volume assessed by bioelectrical impedance (BIA) | 6 weeks on PD and 18 weeks on PD
  Bioelectrical impedance directly measures extracellular fluid volume and total body water. The test is based on the ability to detect differences in the conductive properties of a cell by measuring its resistance (impedance) to electrical current. The technique is reliable for tracking sequential changes in extracellular fluid volume.
Changes in heart rate variability | 6 weeks on PD and 18 weeks on PD
  During the microneurography testing, EKG is recorded. Heart rate and heart rate variability(HRV) will be analyzed from EKG data at baseline, 6 weeks and 18 weeks after starting dialysis.
Changes in central intravascular volume assessed by cardiac ultrasound | 6 weeks on PD and 18 weeks on PD
  Central intravascular volume will be assessed by measuring inferior vena cava (IVC) diameter during cardiac ultrasound at baseline, 6 weeks and 18 weeks on dialysis treatment
Changes in plasma catecholamines levels | 6 weeks on PD and 18 weeks on PD
  *Plasma catecholamines (epinephrine and norepinephrine) increase on a glucose-based peritoneal dialysis regimen and may decrease by adding non-glucose-based solution to the dialysis regimen
Changes in BNP (Brain Natriuretic Peptide)levels | 6 weeks on PD and 18 weeks on PD
  *Brain Natriuretic Peptide (BNP)increases on a glucose-based peritoneal dialysis regimen and may decrease by adding non-glucose-based solution to the dialysis regimen
Changes in plasma insulin levels | 6 weeks on PD and 18 weeks on PD
  *Plasma insulin increases on a glucose-based peritoneal dialysis regimen and may decrease by adding non-glucose-based solution to the dialysis regimen

CONTACTS AND LOCATIONS:
Overall Officials: Marcel Ruzicka, MD, PhD, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- Ottawa Hospital Research Institute, Ottawa, Ontario, Canada